CLINICAL TRIAL: NCT02827474
Title: Perspectives on a Quality Abortion Care Experience: A Patient Centered Approach
Brief Title: We Experience: Perspectives on a Quality Abortion Care Experience: A Patient Centered Approach
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Brenda Pereda, Assistant Professor, University of New Mexico
Other Study IDs: UNMHSC- 16-111
Record Dates: First submitted 2016-07-01; First posted 2016-07-11 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy Termination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (2):
- Patient Participants: Patient participants will participate in two patient interviews.
  Interventions: Other: Patient Interview
- Physician Participants: Provider participants will participate in one provider interview.
  Interventions: Other: Provider Interview

INTERVENTIONS:
Other: Patient Interview — Patient intervention includes a 30 minute interview prior to their abortion procedure and a follow up phone-interview that will be 10-minutes and held 24-72 hours from the procedure.
  Groups: Patient Participants
Other: Provider Interview — For physician participants, providers will be interviewed after completion of the patient's visit and this will be 10-15 minutes.
  Groups: Physician Participants

SUMMARY:
The purpose of this study is to determine aspects of abortion care most important to the patient in creating a "high quality" abortion experience, to investigate patients' expectations of abortion care, and to explore provider perceptions of patients' abortion experiences and assess concordance with patients' perspectives.

DETAILED DESCRIPTION:
The purpose of this study is to determine aspects of abortion care most important to the patient in creating a "high quality" abortion experience, to investigate patients' expectations of abortion care, and to explore provider perceptions of patients' abortion experiences and assess concordance with patients' perspectives.

The investigators will conduct semi-structured interviews with patient participants and providers separately to determine patients' expectations of abortion care as well as the most important aspects of the abortion experience and to explore providers' perceptions of their patients' abortion experience and assess concordance.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting to the Center for Reproductive Health (CRH) for induced abortion for an undesired pregnancy in the first trimester < 14 weeks.
* Women ages 18-45 years.
* Woman must have a completed surgical abortion procedure
* Women must be able to speak English or Spanish.

Exclusion Criteria:

* Women who are unable or unwilling to consent for the study or are unable or unwilling to complete a follow-up interview
* Women who are unable to consent and/or are cognitively impaired.
* Women who are under the age of 18
* Women who are incarcerated.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient Participants: Women presenting to Center for Reproductive Health (CRH) for induced abortion for an undesired pregnancy in the first trimester < 14 weeks and age 18-45 years. Woman must have a completed surgical abortion procedure and be able to speak English or Spanish.
  Provider Participants: Providers must be performing procedures on the day patient participants are recruited and must be willing to give their perspective on the participating patients' abortion experience.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Patient Experience, semi-structured interviews | One year
  The investigators will use semi-structured interviews to determine aspects of abortion care most important to the patients in creating a "high quality" abortion experience.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Pereda, MD, Principal Investigator — University on New Mexico
Locations (1):
- Center for Reproductive Health, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No